CLINICAL TRIAL: NCT03637153
Title: Acute Exposure to Hypoxia in Precapillary Pulmonary Hypertension: Physiological and Clinical Effects at Rest and During Exercise
Brief Title: Acute Exposure to High Altitude on Exercise Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2018-00455_B1
Record Dates: First submitted 2018-07-09; First posted 2018-08-17 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Hypertension
Keywords: exercise capacity; High Altitude; contant loaded exercise test
MeSH Terms: conditions — Hypertension, Pulmonary; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Including a baseline assessment and assessments at Low altitude and High altitude
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Order A (Experimental): Firstly, the participants will have their assessments at low altitude (Low altitude: 470m above sea level) in Zurich and consecutively the exposure to High Altitude (Säntis; 2500m above sea Level).
  Interventions: Other: Assessment at Low Altitude (470m above sea level); Other: Exposure to High Altitude (2500m above sea level)
- Order B (Experimental): Firstly, the participants will exposed to High Altitude (Säntis; 2500m above sea level) and consecutively will they have assessement in Zurich (Low altitude; 470m above sea level).
  Interventions: Other: Assessment at Low Altitude (470m above sea level); Other: Exposure to High Altitude (2500m above sea level)

INTERVENTIONS:
Other: Assessment at Low Altitude (470m above sea level) — Assessment at Low Altitude (in Zurich; 470m above sea level) in order to compare this data with High altitude exposure
Other: Exposure to High Altitude (2500m above sea level) — Exposure to High Altitude (Säntis; 2500m above sea level) for approximately 5 hours

SUMMARY:
Randomized crossover Trial in patients with Pulmonary Hypertension (PAH, CTEPH) to assess the acute response to High Altitude (2500m above sea level) in constant loaded exercise capacity.

DETAILED DESCRIPTION:
Low altitude baseline measurements will be performed in Zurich (460m asl) including Echocardiography, Right heart catheterization, 6MWT, pulmonary function test, clinical assessment and blood gas Analysis.

Randomly assigned to the order of testing, the participants will be tested in Low Altitude (Zurich, 470m) and at High Altitude (2500m).

Towards the end of the exposure after approximately 4 hours, the participants will perform a constant loaded exercise test on an Ergometer with a calculated resistance of their 60% max Workload.

The patients will be encouraged to perform these tests up to their physical exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* PH diagnosed according to internation Guidelines: mPAP ≥ 25 mmHg along with a PAWP ≤15 mmHg during right heart catheterization at the time of Initial diagnosis
* PH class 1 (PAH) or 4 (CTEPH)
* Stable condition, on the same medication for > 4 weeks
* Patient live permanently at an altitude < 1000m asl.

Exclusion Criteria:

* Resting PaO2 ≤7.3 kPA corresponding to the requirement of long-term oxygen therapy > 16hour daily (nocturnal oxygen therapy alone is allowed)
* Severe daytime hypercapnia (pCO2 > 6.5 kPa)
* Susceptibility to high altitude related diseases (AMS, HAPE, etc.) based on previous experienced discomfort at altitudes.
* Exposure to an altitude >1500m for ≥3 nights during the last 4 weeks before the study participation
* Residence > 1000m above sea level
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurological or orthopedic problems with Walking disability
* Women who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
endurance time at High Altitude | 1 day at altitude
  The time of a constant loaded exercise test by an ergometer in sitting position at High Altitude will be compared with the same test at low altitude (370m above sea level)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof., Principal Investigator — University of Zurich
Locations (1):
- Respiratory Clinic, University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Schneider SR, Lichtblau M, Furian M, Mayer LC, Berlier C, Muller J, Saxer S, Schwarz EI, Bloch KE, Ulrich S. Cardiorespiratory Adaptation to Short-Term Exposure to Altitude vs. Normobaric Hypoxia in Patients with Pulmonary Hypertension. J Clin Med. 2022 May 14;11(10):2769. doi: 10.3390/jcm11102769. PMID 35628896